CLINICAL TRIAL: NCT00936221
Title: A Phase II, Double-blind, Randomised Study to Assess the Efficacy of AZD6244 in Combination With Dacarbazine Compared With Dacarbazine Alone in First Line Patients With BRAF Mutation Positive Advanced Cutaneous or Unknown Primary Melanoma
Brief Title: Comparison of AZD6244 in Combination With Dacarbazine Versus (vs) Dacarbazine Alone in BRAF Mutation Positive Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1532C00006
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Melanoma
Keywords: BRAF mutation positive; advanced melanoma; Advanced cutaneous melanoma; Unknown primary melanoma
MeSH Terms: conditions — Melanoma | interventions — AZD 6244; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): AZD6244 in combination with dacarbazine
  Interventions: Drug: AZD6244; Drug: Dacarbazine
- 2 (Placebo Comparator): Placebo in combination with dacarbazine
  Interventions: Drug: Dacarbazine; Drug: Placebo

INTERVENTIONS:
Drug: AZD6244 — oral capsules, 75mg twice daily
  Other Names: selumetinib
  Arms: 1
Drug: Dacarbazine — 1000 mg/m2 iv infusion over at least 60 min. on day 1 of each 21 cycle
  Other Names: DTIC
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
To assess the efficacy in terms of overall survival of AZD6244 in combination with dacarbazine, compared with dacarbazine alone, in first line patients with BRAF mutation positive advanced cutaneous or unknown primary melanoma

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of advanced (inoperable stage III and stage IV) cutaneous or unknown primary melanoma
* Tumor sample confirmed as BRAF mutation positive

Exclusion Criteria:

* Diagnosis of uveal or mucosal melanoma
* Any prior Investigational therapy comprising inhibitors of Ras, Raf or MEK
* Having received an investigational drug within 30 days of starting treatment, or have not recovered from side effects of an investigational drug

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Middleton, Dr, Principal Investigator — Churchil Hospital, Oxford, UK; Caroline Robert, Dr, Principal Investigator — Institute Gustave Roussy, France; Ian Smith, Dr, Study Director — AstraZeneca, Alderley Park, UK
Locations (38):
- United States (2):
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Ijuí
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Czechia (3):
  - Research Site, Brno
  - Research Site, Nový Jičín
  - Research Site, Prague
- France (3):
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Tübingen
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Székesfehérvár
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
- Research Site, Oslo, Norway
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Houston
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
- Research Site, Zurich, Switzerland
- United Kingdom (7):
  - Research Site, Cambridge
  - Research Site, Chelmsford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Oxford
  - Research Site, Sutton

REFERENCES:
- [Derived] Robert C, Dummer R, Gutzmer R, Lorigan P, Kim KB, Nyakas M, Arance A, Liszkay G, Schadendorf D, Cantarini M, Spencer S, Middleton MR. Selumetinib plus dacarbazine versus placebo plus dacarbazine as first-line treatment for BRAF-mutant metastatic melanoma: a phase 2 double-blind randomised study. Lancet Oncol. 2013 Jul;14(8):733-40. doi: 10.1016/S1470-2045(13)70237-7. Epub 2013 Jun 2. PMID 23735514
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=195&filename=CSP-D1532C00006.pdf
- See also: D1532C00006.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=195&filename=D1532C00006.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Selumetinib 75mg BD +Dacarbazine: selumetinib 75mg twice daily + Dacarbazine
- Placebo BD + Dacarbazine: Placebo twice daily + Dacarbazine
Period: Overall Study
Arm/Group | Selumetinib 75mg BD +Dacarbazine | Placebo BD + Dacarbazine
Started | 45 | 46
Received Treatment | 44 | 45
Completed | 44 (13 patients ongoing cutoff + 31 patients who had died.) | 45 (10 patients ongoing at data cutoff + 35 patients who had died.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selumetinib 75mg BD +Dacarbazine | Placebo BD + Dacarbazine | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (14.89) | 51.6 (16.21) | 53.6 (15.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 22 | 28 | 50

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Following progression survival data was collected until documentation of death, withdrawal of consent, loss to follow-up or the final data cut-off, whichever occurred first.
Time Frame: From date of randomization until death, withdrawal of consent or the end of the study. The end of the study was defined as the date all AZD6244 patients had been followed for a minimum of 12 months, or the date of final analysis, whichever was later
Population: Intention to Treat (ITT)
Measure: Median (Full Range); unit: Days
Groups:
- Selumetinib 75mg BD + Dacarbazine: selumetinib 75mg twice daily + dacarbazine
- Placebo + Dacarbazine: Matched Placebo + dacarbazine
Arm/Group | Selumetinib 75mg BD + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 45 | 46
Days | 424 [63 to 760] | 321 [66 to 739]
Statistical Analysis 1: Comparison: Selumetinib 75mg BD + Dacarbazine vs Placebo + Dacarbazine; If the true hazard ratio (HR) is 0.57, 58 deaths provides at least 80% power to demonstrate a statistically significant difference for OS, assuming a 1-sided 10% significance level; Test type: Superiority or Other; p = 0.3873, Regression, Cox — 1-sided p-value; Cox model adjusting for treatment, WHO performance status, LDH, M status and tumour sub-type; Hazard Ratio (HR) = 0.93, 80% CI 2-sided [0.67 to 1.28]

2. Secondary Outcome: Progression Free Survival
Description: PFS is the time from randomisation until the date of objective disease progression as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) or death (by any cause in the absence of progression). Progression is defined using RECIST (v1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: From randomization until evidence of RECIST-defined objective disease progression or data cut off, for a minimum of 12 months since start of treatment
Population: Intention to Treat (ITT)
Measure: Median (Full Range); unit: Days
Arm/Group | Selumetinib 75mg BD + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 45 | 46
Days | 169 [37 to 596] | 92 [32 to 660]

3. Secondary Outcome: Objective Response Rate
Description: ORR rate is defined as the number (%) of subjects with at least one visit response of Complete Response (CR) or Partial Response (PR) , as defined by Response Evaluation Criteria in Solid Tumours (RECIST v1.1) for target lesions and assessed by CT or MRI. CR, Disappearance of all target lesions; PR, ≥30% decrease in the sum of the longest diameter of target lesions. Data obtained up until progression, or last evaluable assessment in the absence of progression, was included in the assessment of ORR
Time Frame: as for outcome 2
Population: Intention to Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Selumetinib 75mg BD + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 45 | 46
Participants
  Response | 18 | 12
  Complete Response | 1 | 1
  Partial Response | 17 | 11
  Non-response | 27 | 34
  Stable Disease >=6 weeks | 13 | 10
  Progression | 14 | 24

4. Secondary Outcome: Change in Target Lesion Tumour Size at Week 12
Time Frame: randomization to week 12
Population: Intention to Treat (ITT)
Measure: Median (Full Range); unit: % change
Arm/Group | Selumetinib 75mg BD + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 45 | 46
% change | -8.85 [-65.22 to 121.77] | 0.22 [-72.50 to 295.79]

ADVERSE EVENTS:
Arm/Group | Selumetinib 75mg BD +Dacarbazine | Placebo BD + Dacarbazine
Serious Adverse Events (participants affected / at risk) | 22/44 | 8/45
Other Adverse Events (participants affected / at risk) | 44/44 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib 75mg BD +Dacarbazine (N=44) | Placebo BD + Dacarbazine (N=45)
Erysipelas (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Left atrial dilatation (Cardiac disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selumetinib 75mg BD +Dacarbazine (N=44) | Placebo BD + Dacarbazine (N=45)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 7 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 6
EYELID OEDEMA (Eye disorders) | 3 | 0
PERIORBITAL OEDEMA (Eye disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 9 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 12 | 13
DIARRHOEA (Gastrointestinal disorders) | 21 | 13
DRY MOUTH (Gastrointestinal disorders) | 6 | 0
DYSPEPSIA (Gastrointestinal disorders) | 6 | 2
FLATULENCE (Gastrointestinal disorders) | 1 | 5
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 0
NAUSEA (Gastrointestinal disorders) | 28 | 25
STOMATITIS (Gastrointestinal disorders) | 8 | 5
VOMITING (Gastrointestinal disorders) | 20 | 14
ASTHENIA (General disorders) | 12 | 5
CHILLS (General disorders) | 3 | 1
FACE OEDEMA (General disorders) | 3 | 1
FATIGUE (General disorders) | 16 | 15
GENERALISED OEDEMA (General disorders) | 6 | 2
LOCALISED OEDEMA (General disorders) | 3 | 0
OEDEMA PERIPHERAL (General disorders) | 19 | 3
PYREXIA (General disorders) | 5 | 5
FOLLICULITIS (Infections and infestations) | 5 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 6
PARONYCHIA (Infections and infestations) | 6 | 0
RASH PUSTULAR (Infections and infestations) | 6 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 2
URINARY TRACT INFECTION (Infections and infestations) | 5 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 | 1
BLOOD CREATININE PHOSPHOKINASE INCREASED (Investigations) | 7 | 0
BLOOD PRESSURE INCREASED (Investigations) | 4 | 0
WEIGHT INCREASED (Investigations) | 3 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 | 11
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 4
DIZZINESS (Nervous system disorders) | 6 | 2
DYSGEUSIA (Nervous system disorders) | 4 | 4
HEADACHE (Nervous system disorders) | 5 | 12
LETHARGY (Nervous system disorders) | 2 | 4
PARAESTHESIA (Nervous system disorders) | 3 | 4
SYNCOPE (Nervous system disorders) | 4 | 0
ANXIETY (Psychiatric disorders) | 5 | 5
BRADYPHRENIA (Psychiatric disorders) | 0 | 3
DEPRESSION (Psychiatric disorders) | 3 | 2
INSOMNIA (Psychiatric disorders) | 3 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 8 | 6
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 23 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 5 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 3 | 1
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 4 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 | 4
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 5 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 2
SKIN CHAPPED (Skin and subcutaneous tissue disorders) | 4 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 3 | 0
HYPERTENSION (Vascular disorders) | 8 | 1
LYMPHOEDEMA (Vascular disorders) | 11 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No